CLINICAL TRIAL: NCT06462482
Title: Peri-Operative Testosterone Administration in Primary Hip Arthroscopy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: American Hip Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHI-004
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Femoro Acetabular Impingement
Keywords: Testosterone; Hypogonadism; Hip arthroscopy
MeSH Terms: conditions — Femoracetabular Impingement; Hypogonadism | interventions — Nandrolone Decanoate; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone Arm (Experimental): The testosterone group will receive a 200mg dose of intramuscular testosterone cypionate (also known as Nandrolone) weekly for 8 weeks beginning 2 weeks prior to surgery.
  Interventions: Drug: Nandrolone Decanoate
- Saline Arm (Placebo Comparator): The saline group will receive a 200mg dose of intramuscular saline weekly for 8 weeks beginning 2 weeks prior to surgery.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nandrolone Decanoate — Nandrolone will be administered to the testosterone group, specifically a 200mg dose weekly for 8 weeks beginning 2 weeks prior to surgery.
  Arms: Testosterone Arm
Drug: Saline — Saline will be administered to the saline group, specifically a 200mg dose weekly for 8 weeks beginning 2 weeks prior to surgery.
  Arms: Saline Arm

SUMMARY:
It is often observed that patients following hip surgery have a hard time with rehabilitation, as patients commonly lose muscle mass and strength around the surgical site. The goal of this study is to learn if giving patients testosterone around their hip surgery can prevent them from losing muscle mass, as well as to see if it will improve their outcomes after surgery. The main question this study aims to answer is: Will perioperative testosterone administration increase lean mass in addition to improving functional and clinical patient reported outcomes greater than placebo?

Researchers will compare patients who were administered testosterone to standard of care (no administration of testosterone) to see if there is a difference in their recovery and outcomes.

Participants will be given either testosterone or saline for eight weeks beginning two weeks prior to surgery. Participants will have to answer questionnaires on how they are doing, as well as will do other testing during this time.

DETAILED DESCRIPTION:
The purpose of this double blinded, randomized controlled trial is to determine if weekly intramuscular testosterone administration can prevent short-term catabolic loss of lean mass in patients undergoing hip arthroscopy and labral repair in addition to improving functional and patient-reported outcome scores. It is hypothesized that perioperative testosterone administration will increase lean mass in addition to improving functional and clinical patient reported outcomes greater than placebo. This is the first study, to our knowledge, investigating the effects of perioperative testosterone administration on male patients undergoing hip arthroscopy and labral repair.

Participants will be randomly assigned to receive testosterone or placebo treatment. This will be performed using a simple 1:1 randomization and will be provided to the study's designated team member who is not associated with the study, to be referred to as the pharmacist. Except for the statistician performing the randomization and the pharmacist, all individuals involved - including the investigators, study team, surgeon, physical therapist, and patient - will be blinded to the assigned treatment.

Informed consent documentation will include an in-depth discussion of the possible, but uncommon, risks of testosterone including allergic reactions, liver function test alterations, breast tenderness, hair growth or loss, polycythemia, and mood or mental changes. These potential adverse events will be monitored during all study visits.

The testosterone group will receive a 200mg dose of intramuscular testosterone cypionate (also known as Nandrolone) weekly for 8 weeks beginning 2 weeks prior to surgery. The 200 mg per week regimen is being selected with the goal of being a dose sufficient to provide an anabolic stimulus, and low enough to minimize potential adverse effects [10-13]. Control participants in the placebo group will follow the same schedule of injections with an intramuscular dose of saline instead of testosterone. All participants will follow a structured, standard of care, rehabilitation protocol within one week of surgery. Common markers of endocrine function will be monitored for potential systemic side effects of testosterone using blood analysis of pituitary hormones including luteinizing hormone (LH) and follicle stimulating hormone (FSH), prostate-specific antigen (PSA), alanine aminotransferase (ALT), hematocrit, hemoglobin, and white blood cell at 2 weeks preoperatively, the day of surgery, and then 2 weeks, 6 weeks, 3 months, and 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Male patients over the age of 18 with a diagnosis of femoroacetabular impingement (FAI) with labral tear will be recruited to the study and screened for eligibility. Inclusion criteria include clinical diagnosis of FAI, age 18 and older, and hypogonadism, defined as a testosterone level <300ng/dL.

Exclusion Criteria:

* . Major exclusion criteria include previous surgery to the affected hip or spine, LCEA < 18, a past medical history significant for allergy to testosterone, prostate cancer, PSA > 4 ng/ml, breast cancer, polycythemia, diabetes mellitus with a HbA1c > 7, BMI < 18 or > 40, and preoperative motion or strength limitations that will affect postoperative rehabilitation.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
modified Harris Hip Score | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome

SECONDARY OUTCOMES:
Total lean body mass | 2 years
  Measuring total lean body mass via Lunar IDXA
Nonarthritic Hip Score | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
HOS-SSS | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
iHOT-12 | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
Age | Before surgery
  Demographic information
Body mass index | Before surgery
  Demographic information
Sex | Before surgery
  Demographic information

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck EC, Nwachukwu BU, Krivicich LM, Malloy P, Suppauksorn S, Jan K, Nho SJ. Preoperative Hip Extension Strength Is an Independent Predictor of Achieving Clinically Significant Outcomes After Hip Arthroscopy for Femoroacetabular Impingement Syndrome. Sports Health. 2020 Jul/Aug;12(4):361-372. doi: 10.1177/1941738120910134. Epub 2020 May 11. PMID 32392094
- [Background] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177
- [Background] Chen F, Lam R, Shaywitz D, Hendrickson RC, Opiteck GJ, Wishengrad D, Liaw A, Song Q, Stewart AJ, Cummings CE, Beals C, Yarasheski KE, Reicin A, Ruddy M, Hu X, Yates NA, Menetski J, Herman GA. Evaluation of early biomarkers of muscle anabolic response to testosterone. J Cachexia Sarcopenia Muscle. 2011 Mar;2(1):45-56. doi: 10.1007/s13539-011-0021-y. Epub 2011 Feb 26. PMID 21475673
- [Background] Serra C, Bhasin S, Tangherlini F, Barton ER, Ganno M, Zhang A, Shansky J, Vandenburgh HH, Travison TG, Jasuja R, Morris C. The role of GH and IGF-I in mediating anabolic effects of testosterone on androgen-responsive muscle. Endocrinology. 2011 Jan;152(1):193-206. doi: 10.1210/en.2010-0802. Epub 2010 Nov 17. PMID 21084444
- [Background] White JP, Baltgalvis KA, Sato S, Wilson LB, Carson JA. Effect of nandrolone decanoate administration on recovery from bupivacaine-induced muscle injury. J Appl Physiol (1985). 2009 Nov;107(5):1420-30. doi: 10.1152/japplphysiol.00668.2009. Epub 2009 Sep 10. PMID 19745189
- [Background] Wu B, Lorezanza D, Badash I, Berger M, Lane C, Sum JC, Hatch GF 3rd, Schroeder ET. Perioperative Testosterone Supplementation Increases Lean Mass in Healthy Men Undergoing Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Orthop J Sports Med. 2017 Aug 9;5(8):2325967117722794. doi: 10.1177/2325967117722794. eCollection 2017 Aug. PMID 28840147
- [Background] Amory JK, Chansky HA, Chansky KL, Camuso MR, Hoey CT, Anawalt BD, Matsumoto AM, Bremner WJ. Preoperative supraphysiological testosterone in older men undergoing knee replacement surgery. J Am Geriatr Soc. 2002 Oct;50(10):1698-701. doi: 10.1046/j.1532-5415.2002.50462.x. PMID 12366624
- [Background] Bhasin S, Storer TW, Berman N, Callegari C, Clevenger B, Phillips J, Bunnell TJ, Tricker R, Shirazi A, Casaburi R. The effects of supraphysiologic doses of testosterone on muscle size and strength in normal men. N Engl J Med. 1996 Jul 4;335(1):1-7. doi: 10.1056/NEJM199607043350101. PMID 8637535
- [Background] Sattler FR, Castaneda-Sceppa C, Binder EF, Schroeder ET, Wang Y, Bhasin S, Kawakubo M, Stewart Y, Yarasheski KE, Ulloor J, Colletti P, Roubenoff R, Azen SP. Testosterone and growth hormone improve body composition and muscle performance in older men. J Clin Endocrinol Metab. 2009 Jun;94(6):1991-2001. doi: 10.1210/jc.2008-2338. Epub 2009 Mar 17. PMID 19293261
- [Background] Basaria S, Coviello AD, Travison TG, Storer TW, Farwell WR, Jette AM, Eder R, Tennstedt S, Ulloor J, Zhang A, Choong K, Lakshman KM, Mazer NA, Miciek R, Krasnoff J, Elmi A, Knapp PE, Brooks B, Appleman E, Aggarwal S, Bhasin G, Hede-Brierley L, Bhatia A, Collins L, LeBrasseur N, Fiore LD, Bhasin S. Adverse events associated with testosterone administration. N Engl J Med. 2010 Jul 8;363(2):109-22. doi: 10.1056/NEJMoa1000485. Epub 2010 Jun 30. PMID 20592293
- [Background] Basaria S, Wahlstrom JT, Dobs AS. Clinical review 138: Anabolic-androgenic steroid therapy in the treatment of chronic diseases. J Clin Endocrinol Metab. 2001 Nov;86(11):5108-17. doi: 10.1210/jcem.86.11.7983. PMID 11701661
- [Background] Bhasin S, Storer TW, Javanbakht M, Berman N, Yarasheski KE, Phillips J, Dike M, Sinha-Hikim I, Shen R, Hays RD, Beall G. Testosterone replacement and resistance exercise in HIV-infected men with weight loss and low testosterone levels. JAMA. 2000 Feb 9;283(6):763-70. doi: 10.1001/jama.283.6.763. PMID 10683055
- [Background] Bhasin S, Woodhouse L, Casaburi R, Singh AB, Bhasin D, Berman N, Chen X, Yarasheski KE, Magliano L, Dzekov C, Dzekov J, Bross R, Phillips J, Sinha-Hikim I, Shen R, Storer TW. Testosterone dose-response relationships in healthy young men. Am J Physiol Endocrinol Metab. 2001 Dec;281(6):E1172-81. doi: 10.1152/ajpendo.2001.281.6.E1172. PMID 11701431
- [Background] Rothney MP, Martin FP, Xia Y, Beaumont M, Davis C, Ergun D, Fay L, Ginty F, Kochhar S, Wacker W, Rezzi S. Precision of GE Lunar iDXA for the measurement of total and regional body composition in nonobese adults. J Clin Densitom. 2012 Oct-Dec;15(4):399-404. doi: 10.1016/j.jocd.2012.02.009. Epub 2012 Apr 26. PMID 22542222